CLINICAL TRIAL: NCT06483321
Title: Effect of Creatine Supplementation on Physical Performance and Body Composition in Vegan Subjects
Brief Title: Effect of Creatine Supplementation on Physical Performance in Vegan Subjects
Acronym: CREATINVEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/2024
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Deficiency; Diet
Keywords: Performance; Vegan diet; Creatine; Strenght
MeSH Terms: conditions — Malnutrition | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine Supplementation (Experimental): Normocaloric vegan diet supplemented with 0.1 g/kg/day of creatine monohydrate
  Interventions: Dietary Supplement: Creatine Supplementation
- Placebo (Placebo Comparator): Normocaloric vegan diet supplemented with 0.1 g/kg/day of placebo (maltodextrin)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine Supplementation — Normocaloric vegan diet supplemented with 0.1 g/kg/day of creatine monohydrate
  Normocaloric diet based solely on foods of plant sources with creatine supplementatio (0.1 g/kg/day)
  Arms: Creatine Supplementation
Dietary Supplement: Placebo — Normocaloric vegan diet supplemented with 0.1 g/kg/day of placebo (maltodextrin)
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the effect of creatine monohydrate supplementation on body composition, physical performance, and muscle creatine levels in vegan individuals over four weeks.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical study aims to evaluate the effect of creatine monohydrate supplementation on body composition, physical performance, and plasma biomarkers in 20 vegan individuals (10 men and 10 women) over a 4-week period. Participants, who will have followed a strict vegan diet for at least 6 months prior to the study's start, will be randomly assigned to one of two groups: one receiving 0.01 grams of creatine monohydrate daily and the other receiving a placebo (maltodextrin). A dietitian-nutritionist will standardize the participants' diet to ensure it is normocaloric and equivalent in macronutrient distribution. To ensure proper dietary control, 3-day dietary records (two weekdays and one weekend day) will be maintained both at the start of the study and during the last week of the intervention.

Assessments will be conducted before the start of the study (week 0) and at the end (week 4), and will include body composition measurements using the InBody system, physical tests (30-meter sprint, dynamometry, countermovement jump (CMJ), maximum isometric force, and a 15-repeated-jumps test), as well as blood analyses for creatine, creatinine, and creatine kinase (CK) levels, and urine analyses for creatine excretion. It is expected that creatine supplementation in vegan subjects will significantly increase lean muscle mass, improve physical performance in the mentioned tests, and elevate muscle creatine levels while decreasing markers of muscle damage (CK). Statistical analysis will include a repeated measures ANOVA to evaluate changes in dependent variables between groups over time, with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Vegan diet for at least 6 months prior to the study's start.
* Aged between 18-40 years.
* Physically active according to the recommendations of the World Health Organization (WHO).
* Body Mass Index (BMI) between 18.5-24.9 kg/m2.
* No tobacco use.
* No or low alcohol consumption and no orthopedic limitations that would interfere with the performance of the study tests.

Exclusion Criteria:

* Chronic diseases that impair athletic performance (cardiovascular, metabolic, gastrointestinal, respiratory) within the last six months.
* Musculoskeletal disease within the last six months.
* Creatine supplementation prior to the study's start

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
30-meter sprint | 4 weeks
  Time (in seconds) taken to complete the 30-meter distance
Countermovement jump (CMJ) | 4 weeks
  Force output and calculates jump height based on flight time and take-off velocity
15-repeated-jumps test | 4 weeks
  Height of each individual jump,recorded in centimeters
Body weight | 4 weeks
  Body weight in kg
Lean mass | 4 weeks
  Lean mass in kg

SECONDARY OUTCOMES:
Maximum isometric force | 4 weeks
  Peak force exerted during the test, typically recorded inkilograms-force (kg)
Blood creatine | 4 weeks
  Milligrams of creatine per deciliter of blood (mg/dL) and in micromoles of creatine per liter of blood (micromoles/L)
Blood creatinine | 4 weeks
  Milligrams of creatinine per deciliter of blood (mg/dL) and in micromoles of creatinine per liter of blood (micromoles/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Francisco de Vitoria University, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No